CLINICAL TRIAL: NCT01763424
Title: Evaluation of Topical Nicotinamide in Combination With Calcipotriol Compared With Calcipotriol Alone for the Treatment of Mild to Moderate Psoriasis.
Brief Title: Nicotinamide in the Treatment of Psoriasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Mehdi Khodadadi, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 390134
Record Dates: First submitted 2013-01-05; First posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — calcipotriene; Niacinamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcipotriol (Active Comparator): Patients applied calcipotriol 0.005% (By LEO Pharmaceuticals, Ballerup, Denmark) for lesions of the other side of the body. The patients uses the medications twice daily (in the morning and before sleeping) for 12 weeks; the total doses of medication used not more than 100 gram per week.
  Interventions: Drug: Calcipotriol
- Calcipotriol plus Nicotinamide (Experimental): Patients applied calcipotriol 0.005% and nicotinamide 4% in combination (By LEO Pharmaceuticals, Ballerup, Denmark) for lesions of one side of the body. The patients uses the medications twice daily (in the morning and before sleeping) for 12 weeks; the total doses of medication used not more than 100 gram per week.
  Interventions: Drug: Calcipotriol plus Nicotinamide

INTERVENTIONS:
Drug: Calcipotriol plus Nicotinamide — Patients applied calcipotriol 0.005% and nicotinamide 4% in combination (By LEO Pharmaceuticals, Ballerup, Denmark) for lesions of one side of the body. The patients uses the medications twice daily (in the morning and before sleeping) for 12 weeks; the total doses of medication used not more than 100 gram per week.
  Arms: Calcipotriol plus Nicotinamide
Drug: Calcipotriol — Patients applied calcipotriol 0.005% (By LEO Pharmaceuticals, Ballerup, Denmark) for lesions of the other side of the body. The patients uses the medications twice daily (in the morning and before sleeping) for 12 weeks; the total doses of medication used not more than 100 gram per week.
  Arms: Calcipotriol

SUMMARY:
This study will determine if combination of topical calcipotriol and nicotinamide is more effective than calcipotriol alone in treatment of psoriasis.

DETAILED DESCRIPTION:
Current treatment strategies of psoriasis are not completely satisfactorily. By inhibiting inflammatory cytokines, nicotinamide may enhance the effects of current topical treatments. Preliminary studies have shown that nicotinamide, which is a vitamin B derivative, is effective in the treatment of psoriasis. According to lack of data, we will investigate the beneficial effects of adding nicotinamide to calcipotriol for patients with mild to moderate psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of 18 to 65 years old,
* Mild to moderate psoriasis; patients must have had less than 15% of the involved body surface, symmetrical plaques (bilateral lesions) or two plaques at least 5 cm apart on the same side of the body with plaque size greater than 2 × 2 cm, but smaller than 15 × 15 cm.
* Willingness to participate

Exclusion Criteria:

* Those who used any medication or niacin and multi-vitamins two weeks, or anti-psoriatic systemic drugs or beta-blockers one month prior to the study,
* Pregnant women,
* Those with the history of renal, hematologic, liver and major psychiatric diseases,
* Those with only scalp, nail, flexural, palmoplantar, or pustular psoriasis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Psoriasis severity | Up to 3 months
  Patients are visited by a dermatologist at baseline and then after the first and third month of therapy, and psoriasis severity is evaluated using the modified psoriasis area and severity index.

SECONDARY OUTCOMES:
Patient's satisfaction | After 3 months
  Patient's satisfaction is evaluated at the end of the trial using a 10-point rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Khodadadi, MD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Skin Diseases and Leishmaniasis Research Center, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Levine D, Even-Chen Z, Lipets I, Pritulo OA, Svyatenko TV, Andrashko Y, Lebwohl M, Gottlieb A. Pilot, multicenter, double-blind, randomized placebo-controlled bilateral comparative study of a combination of calcipotriene and nicotinamide for the treatment of psoriasis. J Am Acad Dermatol. 2010 Nov;63(5):775-81. doi: 10.1016/j.jaad.2009.10.016. PMID 20599292